CLINICAL TRIAL: NCT02753075
Title: A Clinical Study Investigating the Efficacy of Two Experimental Oral Rinses in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: A Study in Dentinal Hypersensitivity (DH) Participants to Assess the Efficacy of an Occluding Dentifrice.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204773
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Experimental Oral Rinse 1 (Experimental): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Experimental Oral Rinse 1 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Device: Experimental Oral Rinse 1; Drug: Fluoride toothpaste
- Experimental Oral Rinse 2 (Experimental): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Experimental Oral Rinse 2 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Device: Experimental Oral Rinse 2; Drug: Fluoride toothpaste
- Placebo Oral Rinse (Placebo Comparator): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Placebo Oral Rinse 2 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Other: Placebo Oral Rinse; Drug: Fluoride toothpaste

INTERVENTIONS:
Device: Experimental Oral Rinse 1 — Oral rinse containing 1.5% w/w KOX, 0ppm F, pH 4.5
  Arms: Experimental Oral Rinse 1
Device: Experimental Oral Rinse 2 — Oral rinse containing 2.0% w/w KOX, 45ppm F, pH 4.5
  Arms: Experimental Oral Rinse 2
Other: Placebo Oral Rinse — Oral rinse containing 0% w/w KOX 0ppm F, pH 4.5
  Arms: Placebo Oral Rinse
Drug: Fluoride toothpaste — Oral rinse containing 1000ppm fluoride as sodium monofluorophosphate

SUMMARY:
This study will investigate the longitudinal efficacy of two experimental oral rinses, one containing 1.5% weight/weight (w/w) dipotassium oxalate monohydride (KOX) /0 Parts per Million (ppm fluoride) and the other 2.0% w/w KOX /45ppm fluoride, for the relief of dentinal hypersensitivity (DH), compared to a placebo oral rinse, when used as an adjunct to twice daily brushing with a standard fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good general health with no clinically significant/ relevant abnormalities in medical history or upon oral examination
* Pre-existing self reported and clinically diagnosed tooth sensitivity
* At screening a minimum of 20 natural teeth and at least two accessible, non-adjacent teeth (incisors, canines or pre-molars) preferably in different quadrants with a signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR),tooth with modified gingival index (MGI) score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1 and tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response).
* At baseline, a minimum of 2 non-adjacent accessible teeth (incisors, canines or premolars) with DH (qualifying tactile threshold Yeaple ≤ 20g, Schiff Sensitivity Score ≥ 2)

Exclusion Criteria:

* Participants with a known or suspected intolerance or hypersensitivity to study products
* Presence of chronic debilitating disease which could affect study outcomes
* Any condition which is causing dry mouth
* Use of an oral care product indicated for the relief of dentine hypersensitivity
* Participation in a DH treatment study in the 8 weeks prior to screening
* Taking daily doses of a medication/ treatment which could interfere with perception of pain or is causing dry mouth
* Require antibiotic prophylaxis for dental procedures
* Dental prophylaxis within 4 weeks of screening
* Treatment of periodontal disease within 12 months of screening
* Scaling or root planning within 3 months of screening
* Tooth bleaching within 8 weeks of screening
* Active caries or periodontitis
* Partial dentures, orthodontic appliances or dental implants which could affect study outcomes
* Pregnant and breast-feeding females
* Main Exclusions for Test Teeth: evidence of current or recent caries; treatment of decay within 12 months of screening; teeth with exposed dentine but with deep, defective or facial restorations; teeth used as abutments for fixed or removable partial dentures; teeth with full crowns or veneers, orthodontic bands or cracked enamel; sensitive teeth with contributing aetiologies other than erosion, abrasion or recession

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-09-08; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 283 participants were screened, out of which 240 participants were randomized.
Groups:
- Experimental Oral Rinse 1: Participants were instructed to brush their teeth with fluoride toothpaste for 1 minute (min) and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 milliliter (mL) of Experimental Oral Rinse 1 (1.5% weight by weight [w/w] dipotassium oxalate monohydrate [KOX], 0 parts per million [ppm] fluoride [F]) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
- Experimental Oral Rinse 2: Participants were instructed to brush their teeth with fluoride toothpaste for 1 min and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 mL of Experimental Oral Rinse 2 (2% w/w KOX, 45ppm F) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
- Placebo Oral Rinse: Participants were instructed to brush their teeth with fluoride toothpaste for 1 min and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 mL of Placebo Oral Rinse (0% w/w KOX) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Started | 79 | 80 | 81
Completed | 71 | 77 | 78
Not Completed | 8 | 3 | 3
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 1 | 3
Not completed — Physician Decision | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Oral Rinse 1: Participants were instructed to brush their teeth with fluoride toothpaste for 1 min and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 mL of Experimental Oral Rinse 1 (1.5% w/w KOX, 0 ppm F) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse | Total
Number analyzed (Participants) | 79 | 80 | 81 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (9.00) | 40.0 (9.81) | 40.5 (8.71) | 40.3 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 70 | 209
  Male | 12 | 8 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score of Experimental Oral Rinses 1 and 2 Against a Placebo Oral Rinse at Week 8
Description: The examiner assessed the participant's response to an evaporative air stimulus for each selected two teeth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity.
Time Frame: Baseline, Week 8
Population: Intent-to-treat (ITT) population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 71 | 77 | 78
score on a scale
  At Baseline | 2.53 (0.422) | 2.55 (0.415) | 2.55 (0.416)
  Change from Baseline at Week 8 | -1.19 (1.097) | -1.29 (0.961) | -1.28 (1.031)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.8290, ANCOVA — For the Week 8 comparisons of two Oral Rinses against the Placebo Rinse, Dunnett's multiplicity adjustment is applied; Least Square (LS) mean difference = 0.09, 95% CI 2-sided [-0.289 to 0.461] — From ANCOVA model with treatment as factor and baseline Schiff score as covariate. Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.9993, ANCOVA — For the Week 8 comparisons of two Oral Rinses against the Placebo Rinse, Dunnett's multiplicity adjustment is applied; LS mean difference = -0.01, 95% CI 2-sided [-0.372 to 0.362] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score of Two Experimental Oral Rinses 1 and 2 at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: ITT population included all participants who are randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2
Number analyzed (Participants) | 71 | 77
score on a scale
  At Baseline | 2.53 (0.422) | 2.55 (0.415)
  Change from Baseline at Week 8 | -1.19 (1.097) | -1.29 (0.961)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.5892, ANCOVA; LS mean difference = 0.09, 95% CI 2-sided [-0.242 to 0.424] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Oral Rinse 1: Participants were instructed to brush their teeth with fluoride toothpaste for 1 min and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 mL of Experimental Oral Rinse 1 (1.5% w/w KOX, 0 ppm fluoride F) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 77 | 79 | 79
score on a scale
  At Baseline | 2.54 (0.420) | 2.54 (0.417) | 2.54 (0.417)
  Change from Baseline at Week 4 | -0.71 (0.864) | -0.83 (0.738) | -0.85 (0.825)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.2825, ANCOVA; LS mean difference = 0.14, 95% CI 2-sided [-0.116 to 0.396] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.8448, ANCOVA; LS mean difference = 0.03, 95% CI 2-sided [-0.229 to 0.280] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.3784, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.141 to 0.371] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Tactile Threshold (Gram [g]) of Two Experimental Oral Rinses 1, 2 and a Placebo Oral Rinse at Week 4
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force has reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g. However, in situations where participants did not give a 'yes' response at force of 80g, the tactile threshold was recorded as >80g. For analysis purposes values recorded as >80g were treated as 90g values.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Median (Full Range); unit: g
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 77 | 79 | 79
g
  At Baseline | 10.00 [10.0 to 20.0] | 10.00 [10.0 to 20.0] | 10.00 [10.0 to 20.0]
  Change from Baseline at Week 4 | 15.00 [0.0 to 80.0] | 10.00 [0.0 to 80.0] | 5.00 [0.0 to 80.0]
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.1688, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-10.00 to 0.000] — Median difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment. Median Difference has been calculated from non-parametric Hodges-Lehmann estimations
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.4380, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 0.000] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.5693, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 0.000] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Tactile Threshold (g) of Two Experimental Oral Rinses 1, 2 and a Placebo Oral Rinse at Week 8
Description: as for outcome 4
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Median (Full Range); unit: g
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 71 | 77 | 78
g
  At Baseline | 10.00 (1.187) [10.0 to 20.0] | 10.00 (1.737) [10.0 to 20.0] | 10.00 (1.971) [10.0 to 20.0]
  Change from Baseline at Week 8 | 40.00 (30.932) [0.0 to 80.0] | 40.00 (30.754) [-5.0 to 80.0] | 40.00 (32.873) [0.0 to 80.0]
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7789, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 0.000] — Median difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment. From non-parametric Hodges-Lehmann estimations
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7214, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 0.000] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.8960, Wilcoxon rank sum test — Wilcoxon rank sum test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 5.000] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Visual Rating Scale (VRS) of Two Experimental Oral Rinses 1, 2 and a Placebo Oral Rinse at Week 4
Description: Participants rated the intensity of their response to the evaporative (air) stimulus using a 10 point VRS. The Participants were asked to rate their pain on a scale of 1 (No Pain) to 10 (intense Pain). A reduction in the score is indicative of an improvement in sensitivity.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 77 | 79 | 79
score on a scale
  At Baseline | 6.88 (1.670) | 6.96 (1.472) | 6.72 (1.692)
  Change from Baseline at Week 4 | -1.57 (1.699) | -1.84 (1.698) | -1.97 (1.819)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.0978, ANCOVA; LS mean difference = 0.45, 95% CI 2-sided [-0.084 to 0.987] — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate. Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.4607, ANCOVA; LS mean difference = 0.20, 95% CI 2-sided [-0.333 to 0.732] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.3542, ANCOVA; LS mean difference = 0.25, 95% CI 2-sided [-0.283 to 0.787] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in VRS of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse) at Week 8
Description: Participants rated the intensity of their response to the evaporative (air) stimulus using a 10 point VRS. The Participants were asked to rate their pain on a scale of 1 ("No Pain") to 10 ("Intense Pain"). A reduction in the score is indicative of an improvement in sensitivity.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 71 | 77 | 78
score on a scale
  At Baseline | 6.92 (1.626) | 6.92 (1.471) | 6.72 (1.703)
  Change from Baseline at Week 8 | -2.63 (2.257) | -2.73 (2.096) | -2.54 (2.325)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.9474, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.665 to 0.711] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7987, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.760 to 0.586] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.7525, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.578 to 0.798] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Groups:
- Experimental Oral Rinse 1: Participants were instructed to brush their teeth with fluoride toothpaste for 1 minute (min) and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 milliliter (mL) of Experimental Oral Rinse 1 (1.5% weight by weight [w/w] dipotassium oxalate monohydrate [KOX], 0 parts per million [ppm] fluoride [F], pH 4.5) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
- Experimental Oral Rinse 2: Participants were instructed to brush their teeth with fluoride toothpaste for 1 min and expectorate. They then rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated followed by rinsing with 10 mL of Experimental Oral Rinse 2 (2% w/w KOX, 45ppm F, pH 4.5) for 1 min and expectorated. This regimen was performed twice daily for 8 weeks.
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 10/79 | 8/80 | 2/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Oral Rinse 1 (N=79) | Experimental Oral Rinse 2 (N=80) | Placebo Oral Rinse (N=81)
ORAL DISCOMFORT (Gastrointestinal disorders) | 4 | 2 | 0
DRY MOUTH (Gastrointestinal disorders) | 3 | 2 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 2 | 1 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 2 | 0 | 0
GLOSSODYNIA (Gastrointestinal disorders) | 1 | 3 | 0
LIP EXFOLIATION (Gastrointestinal disorders) | 1 | 0 | 0
LIP SWELLING (Gastrointestinal disorders) | 1 | 0 | 0
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 0 | 0 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 1 | 0
TOOTH DISORDER (Gastrointestinal disorders) | 0 | 1 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.